CLINICAL TRIAL: NCT03120468
Title: Topiramate Augmenting Strategies for the Treatment of Alcohol Use Disorder
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nassima Ait-Daoud Tiouririne (Other)
Responsible Party: Sponsor-Investigator, Nassima Ait-Daoud Tiouririne, Associate Professor, Director of UVA Center for Leading Edge Addiction Research, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19422
Record Dates: First submitted 2017-03-31; First posted 2017-04-19 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Alcoholism
Keywords: alcohol, alcohol dependence, addiction, alcohol use disorder
MeSH Terms: conditions — Alcoholism; Behavior, Addictive | interventions — Topiramate; Acetylcysteine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Topiramate and N-Acetyl Cysteine (Experimental): Drug: Topiramate and N-Acetyl Cysteine Other Name for Topiramate: Topamax
  Interventions: Drug: Topiramate and N-Acetyl Cysteine
- Topiramate and Placebo (Experimental): Drug: Topiramate and Placebo Other Name for Topiramate: Topamax Other Name for Placebo: Sugar Pill
  Interventions: Drug: Topiramate and Placebo

INTERVENTIONS:
Drug: Topiramate and N-Acetyl Cysteine — Topiramate up to 200 mg/day and N-Acetyl Cysteine 600 mg twice a day for 12 weeks
  Other Names: Topamax
  Arms: Topiramate and N-Acetyl Cysteine
Drug: Topiramate and Placebo — Topiramate up to 200 mg/day and Placebo for 12 weeks
  Other Names: Topamax; Sugar Pill
  Arms: Topiramate and Placebo

SUMMARY:
This is a pilot study designed to evaluate the safety, tolerability of Topiramate (TPM) + N-Acetyl Cysteine (NAC) in combination versus Topiramate (TPM) + placebo for the treatment of alcohol use disorder (AUD).

DETAILED DESCRIPTION:
This is a pilot study designed to evaluate the safety, tolerability of Topiramate (TPM) + N-Acetyl Cysteine (NAC) in combination versus Topiramate (TPM) + placebo in 16 subjects enrolled in a 12 week, randomized, double-blind, outpatient trial. Each subject will receive randomly one of the drug combinations for 12 weeks plus medication management.

Primary Aim 1: To evaluate the safety, tolerability of Topiramate (TPM) and N-Acetyl Cysteine (NAC) in combination or Topiramate (TPM) + placebo for the treatment of Alcohol Use Disorder (AUD). This aim will be accomplished by testing the following:

•Hypothesis 1 - The combination of Topiramate (TPM) and N-Acetyl Cysteine (NAC) will be well tolerated by participants as evidenced by less self-report cognitive side effects (word finding difficulties, difficulties with concentration, and confusion).

Secondary Aim 1: The combination of Topiramate (TPM) and N-Acetyl Cysteine (NAC) or Topiramate (TPM) + Placebo will reduce alcohol drinking. This aim will be accomplished by testing the following:

•Hypothesis 2 - The combination of Topiramate (TPM) and N-Acetyl Cysteine (NAC) or Topiramate (TPM) + Placebo will reduced alcohol drinking , as evidenced by a statistically significant reduction in percentage of heavy drinking days (PHDD) as compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Ages 18 and above
* Good physical health
* Current DSM-V diagnosis of alcohol use disorder
* Currently drinking ≥21 alcohol units/week for women and ≥28 alcohol units/week for men on average in the last 28 days prior to screen.
* Be seeking treatment for problems with alcohol
* Be able to take oral medication and be willing to adhere to the medication regimen.
* Be able to verbalize an understanding of the consent form, able to provide written informed consent, verbalize willingness to complete study procedures, able to understand written and oral instructions in English and able to complete the questionnaires required by the protocol.
* Agree to the schedule of visits, verbally acknowledge that s/he will be able to attend each scheduled visit, participate in phone visits and that s/he does not have any already scheduled events or a job that may substantially interfere with study participation.
* Not have any unresolved legal problems that could jeopardize continuation or completion of the study.
* The pregnancy test for females at screen and prior to randomization must be negative. Additionally, women of childbearing potential must be using an acceptable form of contraception. These include: oral contraceptives, hormonal (levonorgestrel) or surgical implants, or barrier plus spermicide.

Exclusion Criteria:

Please contact site for additional information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive side effects | up to13 weeks
  Collection of self-report cognitive side effects

SECONDARY OUTCOMES:
Percent Heavy Drinking Days (PHDD) | up to 13 weeks
  The timeline follow-back (TLFB) method of measuring alcohol consumption will be used for Percent Heavy Drinking Days (PHDD).
Drinks per Drinking Day | up to 13 weeks
  Additional measures of self-reported drinking outcomes
Percentage of Days Abstinent | up to 13 weeks
  Additional measures of self-reported drinking outcomes
Obsessive compulsive drinking scale (OCDS) | up to 16 weeks
  measurement of craving
Drinking Inventory of Consequence (DrInC) scale | DrInC is at screen, weeks 1,5,9, and 13
  measurement of psychosocial consequences of drinking
Clinical Global Improvement (CGI) scale | up to 16 weeks
  Increase in overall clinical improvement

CONTACTS AND LOCATIONS:
Overall Officials: Nassima Ait-Daoud Tiouririne, M.D., Principal Investigator — University of Virginia
Locations (1):
- UVA Center for Leading Edge Addiction Research, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No